CLINICAL TRIAL: NCT00473564
Title: Robotic Assisted Surgery in Upper Aerodigestive Tract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, William Carroll, MD, Professor of Surgery, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F061228004; HNO 0601 (Other: UAB ComprehensiveCancerCenter ClinicalTrialsReviewCommittee)
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Head and Neck Cancer; Oropharyngeal Cancer; Hypopharyngeal Cancer; Upper Aerodigestive Tract Neoplasms
Keywords: Lesions; Biopsy; Surgery
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TORS Candidates (Experimental): Participants who consented to undergo transoral robotic-assisted surgery using the da Vinci® Robotic System
  Interventions: Procedure: da Vinci® Robotic System

INTERVENTIONS:
Procedure: da Vinci® Robotic System — Head and Neck Surgery using the da Vinci® Robotic System

SUMMARY:
To evaluate the use of the daVinci Robotic System for better visibility and access of head and neck lesions and decreased amount of surgery time.

DETAILED DESCRIPTION:
This trial is a single institution non-randomized study to evaluate the efficacy and safety of the da Vinci® Robotic Surgical System. This study will evaluate the use of the daVinci Robotic System for better visibility and access of head and neck lesions and decreased amount of surgery time. This is a robotic system used by surgeons to perform surgery in a less invasive manner.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck lesions requiring surgical resection, biopsy, or invasive treatment;
* Lesion amendable to robotic assisted surgery treatment;
* Age > 19 years;
* Patient must sign informed consent.

Exclusion Criteria:

* Psychological condition that renders the patient unable to understand the informed consent;
* Poor mouth opening, with maximal opening less than 1.5 cm.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2007-02; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Carroll, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Medical Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dean NR, Rosenthal EL, Carroll WR, Kostrzewa JP, Jones VL, Desmond RA, Clemons L, Magnuson JS. Robotic-assisted surgery for primary or recurrent oropharyngeal carcinoma. Arch Otolaryngol Head Neck Surg. 2010 Apr;136(4):380-4. doi: 10.1001/archoto.2010.40. PMID 20403855
- [Derived] Iseli TA, Kulbersh BD, Iseli CE, Carroll WR, Rosenthal EL, Magnuson JS. Functional outcomes after transoral robotic surgery for head and neck cancer. Otolaryngol Head Neck Surg. 2009 Aug;141(2):166-71. doi: 10.1016/j.otohns.2009.05.014. PMID 19643246
- [Derived] Boudreaux BA, Rosenthal EL, Magnuson JS, Newman JR, Desmond RA, Clemons L, Carroll WR. Robot-assisted surgery for upper aerodigestive tract neoplasms. Arch Otolaryngol Head Neck Surg. 2009 Apr;135(4):397-401. doi: 10.1001/archoto.2009.24. PMID 19380364

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TORS Candidates
Started | 170
Completed | 147
Not Completed | 23
Not completed — robot surgery aborted in OR | 23

BASELINE CHARACTERISTICS:
Arm/Group | TORS Candidates
Number analyzed (Participants) | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 113
  >=65 years | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 15
  White | 154
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adequate Exposure and Access to Oropharyngeal and Hypopharyngeal Head and Neck Lesions
Description: Number of participants with adequate exposure and access for use of the da Vinci® Robotic System in oropharyngeal and hypopharyngeal head and neck lesions
Time Frame: Intraoperatively average of 2 hours
Measure: Number; unit: participants
Arm/Group | TORS Candidates
Number analyzed (Participants) | 170
participants
  Number of participants with adequate exposure | 147
  Number of participants without adequate exposure | 23

2. Secondary Outcome: Assessment of Patients Safety by Evaluating the Number of Participants Who Experienced Known Complications From the Use of the da Vinci® Robotic System During Surgery, Experienced a Need for Conversion to Open Surgery or Required Additional Surgery.
Description: Assessment of patient safety evaluating the number of participants who experienced known complications from the use of the da Vinci® Robotic System during surgery, who experienced a need for conversion to open surgery during the procedure, or who required additional surgery for re-excision of the lesion due to positive margins
Time Frame: 3 - 24 months postoperatively
Population: Participants who successfully underwent transoral robotic-assisted surgery using the da Vinci® Robotic System
Measure: Number; unit: participants
Arm/Group | TORS Candidates
Number analyzed (Participants) | 147
participants
  Known complication: oral hemorrhage | 17
  Known complication: injury to perioral structures | 1
  Known complication: airway edema | 14
  Known complication: nerve injury | 1
  Need for conversion to open procedure during surge | 1
  Need for re-exicision due to positive margins | 11

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | TORS Candidates
Serious Adverse Events (participants affected / at risk) | 21/170
Other Adverse Events (participants affected / at risk) | 121/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TORS Candidates (N=170)
aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
dehydration (Metabolism and nutrition disorders) | 5
oral cavity hemorrhage (Gastrointestinal disorders) | 6
diffuse pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1
excessive mucus in throat (Respiratory, thoracic and mediastinal disorders) | 1
ARDS with respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
pneumonia with respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
dysphagia (Gastrointestinal disorders) | 2
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
myocardial infarction (Cardiac disorders) | 1
hip fracture (Musculoskeletal and connective tissue disorders) | 1
neck edema (General disorders) | 1
chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
vomiting (Gastrointestinal disorders) | 1
leukocytosis (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TORS Candidates (N=170)
dysphagia (Gastrointestinal disorders) | 53
hoarseness (Respiratory, thoracic and mediastinal disorders) | 15
oral pain (Gastrointestinal disorders) | 25
oral yeast infection (Infections and infestations) | 10
trismus (Musculoskeletal and connective tissue disorders) | 9
laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No